CLINICAL TRIAL: NCT03748602
Title: Surgical Thoracic Outlet Decompression Versus Conservative Approach for Patients With Neurogenic Thoracic Outlet Syndrome, a Randomized Controlled Trial
Brief Title: Surgical Thoracic Outlet Decompression for Neurogenic Thoracic Outlet Syndrome
Acronym: STOPNTOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Joep Teijink, Professor in vascular surgery, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL63986.100.17
Record Dates: First submitted 2018-10-31; First posted 2018-11-21 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Neurogenic Thoracic Outlet Syndrome
Keywords: thoracic outlet decompression (TOD)
MeSH Terms: conditions — Thoracic Outlet Syndrome

STUDY DESIGN:
Intervention Model Description: All patients diagnosed with NTOS refractory to conservative physiotherapy treatment (based on criteria produced by the reporting standards) and considered to benefit from TOD in a multidisciplinary TOS-consensus group are considered candidates for this study.
  Patients will be randomized into surgery (TOD) versus conservative physiotherapy. The group randomised for conservative physiotherapy will be offered surgical therapy after 3 months if complaints persist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TOD (Experimental): Thoracic Outlet Decompression (TOD)
  Interventions: Procedure: Thoracic outlet decompression
- Conservative therapy (No Intervention): Physiotherapy and pain relief

INTERVENTIONS:
Procedure: Thoracic outlet decompression — TOD consists out of first rib resection with partial scalenectomy and neurolysis. If there are also complaints below the pectoral minor tendon insertion, a pectoral minor tenotomy is performed.
  Arms: TOD

SUMMARY:
This study will determine the value of TOD (first rib resection with partial scalenectomy and neurolysis) on functionality and quality of life for patients with neurogenic thoracic outlet syndrome. This will be done by randomizing patients into surgery or conservative therapy (physiotherapy and pain relief).

DETAILED DESCRIPTION:
Background:

Neurogenic thoracic outlet syndrome (NTOS) is a condition caused by compression and irritation of the brachial plexus serving the upper extremity. NTOS most frequently occurs in relatively young, active and otherwise healthy individuals and can have a tremendous impact on work, social and personal life. The diagnosis and therapy of NTOS still remains disputed. This is partly because diagnosis is largely clinical and subjective in nature, with no definitive (diagnostic) imaging or diagnostic studies available. As a result, disparities in the definition have produced different opinions regarding diagnostic standards for TOS. Furthermore, given the controversy surrounding the definition and diagnosis of TOS, conflict exists regarding the optimal treatment approach for this condition.

Studies in the last years, have shed light on some of the controversies in diagnosing and treating NTOS. Many patients that benefit from thoracic outlet decompression (TOD) do not fit the historical diagnostic criteria. Those patients (up to 90%) with disputed NTOS have shown improvement of symptoms and functionality after TOD surgery.

Recently, several studies have been published about outcome after TOD surgery for NTOS. These large, multicenter studies show a very low complication rate, ranging from 0-2%, with an extremely low risk of nerve injury.

These studies however report on heterogenous populations, diagnosed without any internationally validated diagnostic criteria. They hint beneficial results for TOD in NTOS patients, however the level of evidence they provide is low. Critics have wondered if the improvements - reported in these trials - are attributed to surgery, or are merely due to coincidence, selection bias, conservative treatment or time (rest).

The society of vascular surgery published reporting standards in 2016 to produce consistency in diagnosis, description of treatment and assessment of results to allow more valuable data to be reported. The investigators believe that a randomized controlled trial - using the reporting standards- could demonstrate the actual added value of a TOD (first rib resection with partial scalenectomy and neurolysis).

Objective:

The objective of this study is to determine the value of TOD (first rib resection with partial scalenectomy and neurolysis) on functionality and quality of life. This will be done by randomizing patients who already received conservative physiotherapy into surgery or continued conservative therapy (physiotherapy and pain relief). After 3 months, the patients with continued maximum conservative therapy will be offered surgery as well if complaints persist. The effect of TOD will be examined by following the change in functionality and quality of life compared to conservative physiotherapy. The durability of these effects on functional assessment and quality of life will also be examined by following patients for 5 years.

Study design:

Single center randomized controlled trial

Study population:

All patients diagnosed with NTOS refractory to conservative physiotherapy treatment (based on criteria produced by the reporting standards) and considered to benefit from TOD in a multidisciplinary TOS-consensus group are considered candidates for this study.

Intervention:

Patients will be randomized into surgery (TOD) versus conservative physiotherapy. The group randomised for conservative physiotherapy will be offered surgical therapy after 3 months if complaints persist.

Main study parameters/endpoints:

Primary endpoint is DASH SCORE. This endpoint will be measured with the DASH questionnaire (Disability of the Arm, Shoulder and Hand) Secondary endpoints will be the score on the CBSQ, VAS scale and SF 12. These endpoints will be measured with the CBSQ questionnaire (Cervical-Brachial Symptoms Questionnaire), VAS scale (Visual Analogue Scale for Pain) and SF 12 (Short Form 12 questionnaire)

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

All patients are operated with the same technique and by the same operator. There is a delay of 3 months for half of the subjects (control group), which is relative due to the early operation (in comparison with the existing waiting list for regular TOD of around 3 months) of the group that is randomised for TOD. There is no denial of 'optimal medical treatment' for any of the participating subjects.

ELIGIBILITY:
Inclusion Criteria:

* High suspicion of NTOS with high level of impairment.

  * The decision to refer a patient with NTOS for surgery is placed at the sole authority of the TOS multidisciplinary workgroup. Members of this workgroup are 2 dedicated vascular surgeons, 2 neurologists, 1 orthopedic surgeon, 3 physiotherapists, 2 radiologists, 3 anesthesiologists.
  * This decision is based on the reporting standards published by Illig et al. in 2016. If a patient fits the criteria postulated in the reporting standards and if there is consensus within the multidisciplinary team, only then patients are referred for TOD.
* Fit for surgery, at the discretion of the treating vascular surgeon and anesthesiologist.
* Signed informed consent form.
* 18 years of age or older
* Dutch or English speaking patients

Exclusion Criteria:

* Unfit for surgery, at the discretion of the treating vascular surgeon and anesthesiologist.
* Younger than 18 years of age
* Patients that do not speak Dutch or English.
* Patients with a history of TOD
* Patients that did not receive previous conservative physiotherapy for this condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Disability of the Arm, Shoulder and Hand (DASH) score | Change in this outcome will be measured at 0, 3, 6, 12, 24, 36 and 60 months after inclusion
  This questionnaire is validated for neurogenic thoracic outlet syndrome and was developed by the American Academy of Traumatology. It includes 30 questions related to symptoms of daily activities and social and psychological functions. Scores range from asymptomatic (0) to totally invalid (100).

SECONDARY OUTCOMES:
Chance in Cervical-Brachial Symptoms (CBSQ) Questionnaire score | Change in this outcome will be measured at 0, 3, 6, 12, 24, 36 and 60 months after inclusion
  This questionnaire is validated for neurogenic thoracic outlet syndrome and consist out of 12 questions with the answer going from 0 to 10, 2 questions Y/N answers, 1 question with a visual feedback which parts of the neck, shoulder, arm or hand have most symptoms.
Change in Visual Analogue Scale (VAS) for Pain | Change in this outcome will be measured at 0, 3, 6, 12, 24, 36 and 60 months after inclusion
  This scale measures pain going from 0 (none) to 10 (intens) Patients can chose any number between 0 and 10 to accuratly rate their pain.
Change in Short Form 12 (SF-12) questionnaire score | Change in this outcome will be measured at 0, 3, 6, 12, 24, 36 and 60 months after inclusion
  This questionnaire measures quality of life. It consist out of 12 questions with answers going from Y/N to 0 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Joep Teijink, MD, PhD, Principal Investigator — Vascular surgeon - Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Ziekenhuis, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No